CLINICAL TRIAL: NCT07405762
Title: Mechanisms of Recovery Phenotypes: Early Neurovascular Decoupling Trajectories After Revascularization in Acute Ischemic Stroke Using Multimodal Monitoring
Brief Title: Early Neurovascular Decoupling Trajectories After Revascularization in Acute Ischemic Stroke
Acronym: MAP-END
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20262039; XJLL-KY-20262039 (Other: Xijing Hospital)
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIS Revascularization Cohort: Adult patients diagnosed with acute ischemic stroke (AIS) due to anterior circulation large vessel occlusion, who have undergone successful endovascular thrombectomy (achieving mTICI grade 2b or 3 reperfusion) within 24 hours of symptom onset.
  Interventions: Diagnostic Test: Multimodal Neuromonitoring

INTERVENTIONS:
Diagnostic Test: Multimodal Neuromonitoring — A battery of assessments performed at Days 1-3 and Day 7 post-thrombectomy to evaluate neurovascular decoupling. This includes Transcranial Doppler (TCD) for cerebral hemodynamics, Electroencephalography (EEG) for neural activity, and F-wave studies for spinal motoneuron excitability.

SUMMARY:
Background:

Recanalization therapy is the standard treatment for acute ischemic stroke (AIS), yet patient outcomes remain highly heterogeneous. The underlying mechanisms of this variability are not fully understood. Neurovascular coupling (NVC), the tight link between neural activity and cerebral blood flow, is fundamental for brain function. Its disruption (neurovascular decoupling) after stroke is hypothesized to be a key determinant of recovery, but its dynamic early trajectory and predictive value for long-term functional recovery are poorly characterized.

Purpose:

This observational study aims to delineate the early trajectory of neurovascular decoupling following endovascular thrombectomy in AIS patients and to investigate its association with long-term functional outcome. We seek to construct a single composite biomarker by integrating multimodal data, and to evaluate its predictive value for 90-day recovery.

Methods:

A prospective cohort of AIS patients who undergo successful endovascular thrombectomy will be enrolled. Multimodal monitoring will be performed at specific early time points: within Days 1-3 and at Day 7 post-procedure. Assessments include: Transcranial Doppler (TCD) for cerebral hemodynamics, Electroencephalography (EEG) for neural activity, and F-wave studies for spinal motoneuron excitability. Clinical severity will be assessed using the National Institutes of Health Stroke Scale (NIHSS) concurrently. The primary outcome is the early trajectory of a composite neurovascular decoupling index. The key predictive relationship between this trajectory and 90-day functional status (assessed using the modified Rankin Scale, mRS) will be evaluated.

Significance:

This study will provide novel insights into the early neurophysiological changes following successful thrombectomy. By defining the trajectory of neurovascular decoupling in the critical first week and linking it to long-term function, the findings may contribute to the development of early predictive models and guide personalized rehabilitation strategies.

DETAILED DESCRIPTION:
Study Title:Early Neurovascular Decoupling Trajectories after Revascularization in Acute Ischemic Stroke using Multimodal Monitoring（MAP-END）

1. Background:

   Despite successful revascularization with endovascular thrombectomy (EVT) for acute ischemic stroke (AIS), significant heterogeneity persists in patients' functional recovery. The underlying physiological mechanisms of this variability remain poorly understood, limiting accurate prognosis and the development of personalized rehabilitation strategies.

   Neurovascular coupling (NVC), the precise physiological link between neural activity and regional cerebral blood flow, is fundamental for normal brain function. Post-stroke, factors such as ischemia-reperfusion injury and neuroinflammation may lead to NVC dysfunction, i.e., neurovascular decoupling. This decoupling is hypothesized to be a critical bridge connecting the primary ischemic insult to secondary neurological dysfunction and poor recovery.

   Currently, the dynamic evolution of early neurovascular decoupling (particularly in the hyper-acute to sub-acute phases) following successful thrombectomy in AIS patients is not well characterized. Furthermore, whether such dynamic trajectories are systematically associated with distinct long-term functional recovery phenotypes lacks evidence from multimodal physiological monitoring. This study hypothesizes that quantifiable, heterogeneous trajectories of neurovascular decoupling exist in the early post-thrombectomy period and that these distinct trajectory patterns can predict patients' 90-day functional outcomes.
2. Objectives:

   2.1.Primary Objective: To delineate and quantify the trajectories of early neurovascular decoupling (within Days 1-3 and at Day 7) in AIS patients following successful endovascular thrombectomy.

   2.2.Secondary Objectives: To investigate the association between early neurovascular decoupling trajectories (based on TCD, EEG, and F-wave parameters) and patients' 90-day functional outcome (modified Rankin Scale, mRS).

   To explore differences in clinical characteristics, infarct volume, and collateral circulation among subgroups defined by different neurovascular decoupling trajectories.
3. Study Design:

   A prospective, single-center, observational cohort study.
4. Study Population:

   4.1.Target Population: Adult patients with AIS due to anterior circulation large vessel occlusion who successfully undergo endovascular thrombectomy (mTICI grade 2b-3) within 24 hours of symptom onset.

   4.2.Sample Size: This is an exploratory study. We plan to consecutively enroll all eligible patients over a 24-month period, with a target sample size of approximately 180 participants.
5. Methods:

   5.1.Data Collection Time Points:

   All research-related assessments will be conducted at the following fixed time points:

   T1 (Baseline/Early Phase): Within 24-72 hours post-thrombectomy. T2 (Sub-acute Phase): At Day 7 (±1 day) post-thrombectomy. T3 (Long-term Outcome): At Day 90 (±7 days) post-thrombectomy. 5.2.Assessments and Tools: A. Multimodal Physiological Monitoring - Performed at T1 and T2.

   Transcranial Doppler (TCD):

   Purpose: To assess cerebral hemodynamic status. Parameters: Peak systolic velocity (PSV), end-diastolic velocity (EDV), mean flow velocity (MFV), and pulsatility index (PI) will be measured in bilateral middle cerebral arteries (MCA). The affected-to-unaffected side ratios will be calculated.

   Electroencephalography (EEG):

   Purpose: To assess cortical neuroelectrical activity. Method: Resting-state EEG recordings for at least 30 minutes using the standard 10-20 system.

   Analysis Parameters: Relative power spectral density (δ, θ, α, β bands), brain symmetry indices (e.g., alpha-delta power ratio symmetry), and functional connectivity metrics within specific frequency bands.

   F-wave Studies:

   Purpose: To assess spinal anterior horn motoneuron excitability. Method: Stimulation of the median or ulnar nerve on the affected side (and the unaffected side if feasible).

   Parameters: F-wave persistence, minimal latency, mean latency, and F-wave amplitude/M-wave amplitude ratio.

   B. Clinical Assessments Neurological Deficit: Assessed using the National Institutes of Health Stroke Scale (NIHSS) at T1, T2, and T3.

   Functional Outcome: Assessed at T3 via face-to-face interview or standardized telephone interview using the modified Rankin Scale (mRS). The primary analysis will dichotomize the mRS into favorable outcome (mRS 0-2) and unfavorable outcome (mRS 3-6).

   C. Imaging Data - Collected from clinical records. Baseline Imaging: Stroke etiology (TOAST classification), assessment of infarct core and penumbra (based on CTP or MRI-DWI/PWI).

   Post-thrombectomy Imaging: Final infarct volume (measured on DWI or FLAIR sequences 24-48 hours post-procedure), mTICI grade.

   Vascular Imaging: Collateral circulation grading (based on CTA). 5.3.Key Variables and Definitions Neurovascular Decoupling Trajectory: Will be identified by applying longitudinal data analysis models (e.g., Group-Based Trajectory Modeling) to the composite index derived from TCD mean flow velocity of the middle cerebral artery, EEG power in the C3/C4 electrodes, and F-wave persistence across T1 and T2 time points.
6. Statistical Analysis Plan 6.1.Descriptive Statistics: Baseline demographic, clinical, and imaging characteristics will be reported.

   6.2.Trajectory Modeling: Group-Based Trajectory Modeling (GBTM) or Latent Class Growth Analysis (LCGA) will be used to identify distinct patterns of longitudinal change trajectories in neurovascular parameters from T1 to T2.

   6.3.Association Analysis: Multivariable logistic regression models, adjusted for known prognostic factors (e.g., age, baseline NIHSS, infarct volume, mTICI grade), will be used to test whether membership in a specific identified "neurovascular decoupling trajectory" pattern is independently associated with 90-day favorable/unfunctional outcome.

   6.4.Predictive Performance: The area under the receiver operating characteristic curve (AUC) of a predictive model combining clinical variables and specific neurovascular trajectory patterns will be calculated and compared against a baseline model containing clinical variables only.

   6.5.Subgroup Analysis: Baseline characteristics will be compared among the defined trajectory patterns.

   6.6.Significance Level: A two-sided p-value < 0.05 will be considered statistically significant. Appropriate corrections for multiple comparisons (e.g., Bonferroni) will be applied.
7. Ethical and Regulatory Considerations The study protocol has been reviewed and approved by the Ethics Committee of Xijing Hospital (Approval Number: XJLL-KY-20262039).

   Written informed consent will be obtained from all participating patients or their legally authorized representatives prior to enrollment.

   The study will be conducted in strict accordance with the principles of the Declaration of Helsinki. All collected data will be de-identified, used solely for the purposes of this study, and stored in a secure, encrypted database.
8. Data Sharing Statement De-identified individual participant data, along with the study protocol and statistical analysis plan, will be made available to researchers who provide a methodologically sound proposal after the publication of the primary results. Data sharing requests will be subject to review and approval by the study steering committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years
2. Acute ischemic stroke due to occlusion of the anterior circulation large vessel (terminal internal carotid artery, or M1/M2 segment of the middle cerebral artery), confirmed by computed tomography angiography (CTA) or magnetic resonance angiography (MRA).
3. Underwent endovascular thrombectomy with successful reperfusion, defined as a post-procedural modified Thrombolysis in Cerebral Infarction (mTICI) grade of 2b or 3.
4. Time from symptom onset to femoral artery puncture is ≤ 24 hours.
5. Written informed consent is provided by the patient or their legally authorized representative.

Exclusion Criteria:

1. Pre-stroke disability defined as a modified Rankin Scale (mRS) score ≥ 2.
2. Severe impairment of consciousness within 24 hours post-thrombectomy, defined as a Glasgow Coma Scale (GCS) score ≤ 8.
3. Inadequate temporal bone window preventing acquisition of stable blood flow signals by Transcranial Doppler (TCD).
4. Conditions that may significantly compromise electroencephalography (EEG) quality, such as history of significant traumatic brain injury, skull defect, or intracranial metallic devices.
5. Conditions that may invalidate F-wave studies, including peripheral neuropathy, cervical radiculopathy, or primary disease of the target muscles.
6. Concurrent severe organ failure, malignancy, or a life expectancy of less than 3 months.
7. Pregnancy or lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (aged 18-85) with acute anterior circulation large vessel occlusion stroke, who have undergone successful endovascular thrombectomy within 24 hours of symptom onset, and are able to undergo early multimodal neuromonitoring.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2028-06-05 (Estimated); Study Completion 2028-09-05 (Estimated)

PRIMARY OUTCOMES:
Trajectory of Neurovascular Decoupling Index | From post-thrombectomy Day 1 to Day 7
  The longitudinal change (trajectory) of a composite neurovascular decoupling index from post-thrombectomy Day 1 to Day 7. The index is a single continuous variable calculated by integrating normalized scores from three key modalities: Transcranial Doppler (TCD) mean flow velocity (MFV) of the middle cerebral artery, Electroencephalography (EEG) power in the C3/C4 electrodes (over the sensorimotor cortex), and F-wave persistence. Distinct patterns will be derived from this index trajectory for subsequent analysis.

SECONDARY OUTCOMES:
90-day Functional Outcome | 90 days (± 7 days) post-thrombectomy
  Functional status assessed using the modified Rankin Scale (mRS). The outcome will be analyzed both as an ordinal scale (0-6) and dichotomized into favorable outcome (mRS score 0-2) versus unfavorable outcome (mRS score 3-6).
Early Neurological Deficit Change | From baseline (Days 1-3) to Day 7 post-thrombectomy
  Change in the National Institutes of Health Stroke Scale (NIHSS) score between baseline (post-thrombectomy Days 1-3) and Day 7 post-thrombectomy.
Neurovascular Decoupling Trajectory patterns as a Predictor of 90-day Outcome | At 90 days post-thrombectomy (using data from Days 1-7)
  Discriminative ability (measured by the Area Under the Receiver Operating Characteristic Curve, AUC) for predicting the dichotomized 90-day functional outcome (mRS 0-2 vs 3-6), using the neurovascular decoupling trajectory patterns derived from the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Lang Jin, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in the primary publication (including demographics, clinical scores, multimodal monitoring parameters, and outcomes) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data and supporting documents will become available beginning 6 months after the publication of the primary results manuscript and will remain accessible for at least 5 years. Requests can be submitted during this period.
Access Criteria: Access will be granted to researchers with a methodologically sound proposal for purposes of replicating analyses, conducting individual participant data meta-analysis, or addressing secondary research questions aligned with the original study objectives. Proposals should be submitted directly to the corresponding author (Dr. Lang Jin, silencelang@163.com) and will be reviewed by the study steering committee. Requestors will need to sign a data use/transfer agreement.
URL: https://www.ClinicalTrials.gov